CLINICAL TRIAL: NCT01651013
Title: Multicentered Observational Prospective Cohort Study on the Treatment of Metastatic Colorectal Cancer and the Role of Evaluating K-Ras
Brief Title: Observational Study on Treatment of Metastatic Colorectal Cancer and the Role of K-Ras
Acronym: CALLAS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Other Study IDs: CALLAS
Record Dates: First submitted 2012-07-24; First posted 2012-07-26 (Estimated); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- metastatic colorectal cancer

SUMMARY:
The purpose of this study is to describe the treatments received and outcomes of patients with metastatic colorectal cancer, what percentage of these patients have K-Ras mutation of the tumor, and to describe the costs of treatments. Information will also be collected regarding risk factors, variables among treatment centers and patients, and explorative analyses will be done to try to identify factors that impact prognosis and factors that predict tolerability and response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis colorectal carcinoma
* Metastatic disease
* Signed informed consent

Exclusion Criteria:

* Prior treatment of metastatic colorectal cancer
* Refusal or incapability of providing informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at participating Institutes who are candidate for first-line treatment of metastatic colorectal cancer
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2010-10; Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
percentage of patients enrolled in a clinical trial | two years
percentage of patients who undergo K-Ras mutation study | 2 years
Percentage of patients with K-Ras mutation | 2 years

OTHER OUTCOMES:
metastatic colorectal cancer treatments used in clinical practice, according to participating center | 2 years
patient outcome according to K-Ras status | two years
estimated costs per treatment per center | 2 years
disease outcome per patient per treatment received | 2 years
factors that influence patient prognosis | 2 years
  exploratory analyses
predictive factors for response to treatment | 5 years
  exploratory analyses

CONTACTS AND LOCATIONS:
Overall Officials: R. V. Iaffaioli, M.D., Principal Investigator — National Cancer Institute, Naples; G. Nasti, M.D., Principal Investigator — National Cancer Institute, Naples; M. C. Piccirillo, M.D., Principal Investigator — National Cancer Institute, Naples
Locations (4):
- Italy (4):
  - A.O.G. Rummo, Benevento
  - Istituto Nazionale dei Tumori , Oncologia Medica - Dipartimento Entero-proctologico, Napoli
  - Ospedale Civile Umberto I, Nocera Inferiore
  - C:R.O. Regione Basilicata Ospedale Giustino Fortunato, Rionero in Vulture